CLINICAL TRIAL: NCT04505657
Title: Lidocaine Spray Plus Oral Celecoxib for Pain Control During Hysterosalpingography: a Randomized Controlled Trial
Brief Title: Lidocaine Spray Plus Oral Celecoxib for Pain Control During Hysterosalpingography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aswan University Hospital (Other)
Responsible Party: Principal Investigator, hany farouk, A Professor, Aswan University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: aswu/351/5/19
Record Dates: First submitted 2020-08-06; First posted 2020-08-10 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: IUCD Complication
MeSH Terms: interventions — Celecoxib; Lidocaine

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Who Masked: Participant
Masking Description: randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Celecoxib plus lidocaine (Experimental): Celecoxib 200 mg (Celebrex® 200, Pﬁzer,USA) administered orally 2 h before the procedure +10% lidocaine spray 4 puffs during the procedure
  Interventions: Drug: celecoxib plus lidocaine
- Celecoxib (Active Comparator): Celecoxib 200 mg (Celebrex® 200, Pﬁzer,USA) administered orally 2 h before the procedure +Sterile water 4 puffs during the procedure
  Interventions: Drug: Celecoxib
- lidocaine (Active Comparator): placebo to celecoxib administered orally 2 h before the procedure +10% lidocaine spray 4 puffs during the procedure
  Interventions: Drug: lidocaine

INTERVENTIONS:
Drug: celecoxib plus lidocaine — Celecoxib 200 mg (Celebrex® 200, Pﬁzer,USA) administered orally 2 h before the procedure +10% lidocaine spray 4 puffs during the procedure
  Other Names: experimental
  Arms: Celecoxib plus lidocaine
Drug: Celecoxib — Celecoxib 200 mg (Celebrex® 200, Pﬁzer,USA) administered orally 2 h before the procedure +Sterile water 4 puffs during the procedure
  Other Names: Active Comparator
  Arms: Celecoxib
Drug: lidocaine — placebo to celecoxib administered orally 2 h before the procedure +10% lidocaine spray 4 puffs during the procedure
  Other Names: Active Comparato
  Arms: lidocaine

SUMMARY:
our aims to investigate the effectiveness of10% Lidocaine Spray plus oral celecoxib for Pain Control During Hysterosalpingography

DETAILED DESCRIPTION:
hysterosalpingography can cause pain and discomfort in several ways: Use of the tenaculum to grasp the cervix and straighten the uterus for proper insertion; trans-cervical actions including measuring uterine depth, inserting the cannula; and injection of the dye

ELIGIBILITY:
Inclusion Criteria:

* any patient came for Hysterosalpingography

Exclusion Criteria:

* any patient has contraindication to Hysterosalpingography

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — female request hystrosalpingogram
Enrollment: 150 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-09-27 (Actual)

PRIMARY OUTCOMES:
Mean pain score during the procedure | 10 minuets
  Assessment of pain using visual analog scale 0-10, 0 = minimum and 10 = maximum scores

CONTACTS AND LOCATIONS:
Overall Officials: nahla w Shady, md, Study Chair — Aswan universirty
Locations (1):
- Aswan University Hospital, Aswān, Egypt

IPD SHARING:
Plan to Share IPD: No